CLINICAL TRIAL: NCT00488254
Title: The Long QT Syndrome in Pregnancy
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Roanne Preston, University of British Columbia
Other Study IDs: H06-03385
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Long QT Syndrome
Keywords: Long QT Syndrome; Romano Ward; Jervell-Lange Nielson Syndrome
MeSH Terms: conditions — Long QT Syndrome; Jervell-Lange Nielsen Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Long QT Syndrome (LQTS) is a disease of young adults and can affect women of child bearing age. Suffers of LQTS are at risk of ventricular dysrhythmias including torsades de pointes and ventricular fibrillation.

Pregnancy increases the chance that any mother may have an abnormal heart rhythm or arrhythmia. This chance is higher with the LQTS. There are only a few reported cases of women with the LQTS having a baby in the medical literature. This can make it difficult for the doctor caring for a pregnant woman with the long QT syndrome - especially should they need an anesthetic.

We would like to study as many women who have had a baby who have the long QT syndrome to give us a better idea of whether there are any arrhythmias occurring at the time of delivery.

DETAILED DESCRIPTION:
This will be a retrospective analysis of all LQTS women managed at St. Paul's or BC Women's who have been pregnant in the last 5 years. These two hospitals both have a provincial role in the care of pregnant women, BC Women's as the designated provincial tertiary maternity care referral centre, and St. Paul's through its provincial PATCH clinic. Using the data from these two centres should capture the majority of LQTS cases in parturients in the province. We will search for these women from the Department of Anesthesia BC Women's consult database, the St. Paul's Cardiac Obstetrical Care database, and BC Women's Health Records using International Classification of Diseases - 10 coding for long QT. Then, after obtaining patient consent, review the charts collecting data using the data entry form. The cases will then be compared and any conclusions into the different anesthetic managements made.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with diagnoses of Long QT Syndrome, Romano Ward and Jervell - Lange Nielson Syndrome who delivered at BC Women's Hospital or St Paul's Hospital.

Exclusion Criteria:

* Non consent to participation in the study
* Age less than 19
* Non English speaker

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women managed at St. Paul's or BC Women's, Vancouver, who have been pregnant in the last 5 years
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2007-06; Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roanne Preston, MD, Principal Investigator — University of British Columbia; Elizabeth Drake, MD, Study Director — University of British Columbia; Joanne Douglas, MD, Study Director — University of British Columbia; Marla Kiess, MD, Study Director — University of British Columbia; Stanley Tung, MD, Study Director — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada